CLINICAL TRIAL: NCT04986670
Title: NutriCare Intervention on Optimizing Nutritional Status, Reducing Treatment-Related Toxicities, and Improving Quality of Life Among Vulnerable Patients With Lung Cancer
Brief Title: NutriCare Plus a Medically Tailored Meal Intervention Among Patients With Lung Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: Fox Chase Cancer Center (Other); M.D. Anderson Cancer Center (Other); Ohio State University (Other); Tufts Medical Center (Other)
Responsible Party: Principal Investigator, Fang Fang Zhang, Associate Professor, The Neely Family Professor and Associate Professor, Tufts University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00000203
Record Dates: First submitted 2021-07-13; First posted 2021-08-03 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Lung Cancer, Small Cell; Lung Cancer Metastatic; Lung Cancer Recurrent; Treatment Side Effects; Lung Cancer, Non-small Cell; Nutritional Imbalance
Keywords: lung cancer; malnutrition; vulnerability; medically tailored meals; nutrition counseling
MeSH Terms: conditions — Small Cell Lung Carcinoma; Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Malnutrition | interventions — Nutrition Assessment

STUDY DESIGN:
Intervention Model Description: For the proposed study, we will randomize participants into two groups at a 1:1 ratio to an intervention or an enhanced control group. For participants randomized to the enhanced control group, the NutriTool, the oncology care team will provide participants with a nutrition toolkit involving printed educational materials. For participants randomized to the intervention group, the NutriCare, the oncology care team will additionally provide participants with home-delivery of medically tailored meals and referral to registered dietitians (RDs) for remotely-delivered nutrition counseling.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NutriCare (Experimental): The oncology care team will provide participants with nutrition toolkit involving printed educational materials, a nutrition prescription, referral to registered dietitians (RDs) for remotely-delivered medical nutrition therapy counseling, and home-delivery of medically tailored meals.
  Interventions: Behavioral: Nutritional Counseling; Other: Medically Tailored Meals (MTMs); Behavioral: Nutrition Prescription; Other: Nutrition Assessment; Behavioral: Nutrition Toolkit; Behavioral: Monthly Emails
- NutriTool (Active Comparator): The oncology care team will provide participants with a nutrition toolkit involving printed educational materials.
  Interventions: Behavioral: Nutrition Toolkit; Behavioral: Monthly Emails

INTERVENTIONS:
Behavioral: Nutritional Counseling — Medical oncology providers will refer participants to oncology RDs for remotely delivered medical nutrition therapy counseling. For cohort 1, participants will receive nutrition counseling for 8 months. The counseling will be provided on a weekly basis during the first 6 months and every other week during the last 2 months (for cohort 1 only). For cohort 2, participants will receive nutrition counseling for 6 months. The ultimate frequency of nutrition counseling being provided to each participant will also be adjusted according to the participant's preference and needs.
  Arms: NutriCare
Other: Medically Tailored Meals (MTMs) — Medically tailored meals will be provided to participants in the intervention group for a total of 24 weeks for both cohorts. During the first 8 weeks of the intervention, 3 meals/day will be provided each week for a total of 168 meals per participant. It will be followed by less frequent meal provision during the subsequent 16 weeks following this schedule: 3 meals/day will be provided every other week for the next 8 weeks (a total of 84 meals per participant); and 3 meals/day will be provided every four weeks during the last 8 weeks (a total of 42 meals per participant). The number of meals provided to each participant may be adjusted according to participant's preference and needs.
  Arms: NutriCare
Behavioral: Nutrition Prescription — Oncology providers will advise participants with lung cancer to follow evidence-based nutrition recommendations using a Nutrition Prescription. The Nutrition Prescription aims to enhance providers' role in communicating basic nutrition advice to participants with lung cancer. It contains seven recommendations, adapted from the newly released Cancer Prevention Recommendations by WCRF/AICR with strong evidence-base.
  Arms: NutriCare
Other: Nutrition Assessment — Oncology care providers will assess the nutritional status of patients with lung cancer using PG-SGA Short Form (the Scored Patient-Generated Subjective Global Assessment). PG-SGA is an interdisciplinary patient assessment in oncology and other chronic catabolic conditions. The short form contains four patient generated historical components (weight history, food intake symptoms, and activities and function).
  Arms: NutriCare
Behavioral: Nutrition Toolkit — Patients will receive a printed copy of a Nutrition Toolkit from providers. Evidence-based nutrition recommendations have been compiled for cancer survivors from 4 sources into a Nutrition Toolkit. The sources include: (1) AmericanCancer Society (ACS) Nutrition and Physical Activity Guidelines for Cancer Survivors; (2)World Cancer Research Fund / American Institute for Cancer Research (WFRF/AICR) Cancer Nutrition Guide; (3) National Cancer Institute (NCI) Eating Hints; and (4) National Comprehensive Cancer Network (NCCN) Guidelines for Cancer Survivors. The Nutrition Toolkit outlines topics about the impact of cancer treatment on dietary intake patterns and quality, strategies to manage treatment-related eating issues, maintaining a healthy weight post treatment, and evidence-based recommendations and practical. Nutrition Toolkit strategies for improving diet quality and maintaining an optimal weight for cancer survivors.
Behavioral: Monthly Emails — Monthly emails will be sent to participants to encourage the use of the toolkit with healthy recipes and general nutrition information.

SUMMARY:
The NutriCare study aims to develop, implement, and evaluate the efficacy of an innovative intervention strategy (medically tailored meals plus nutrition counseling) to integrate nutrition into the standard of care for oncology to improve outcomes of vulnerable patients with lung cancer. The NutriCare study evaluates the efficacy of the intervention on optimizing nutritional status, reducing treatment-related toxicities, and improving the quality of life of patients with lung cancer who are economically disadvantaged, uninsured, racial and ethnic minorities, elderly, and/or rural residents from four major medical centers in diverse regions of the United States (U.S.). There will be two cohorts for NutriCare with cohort 1 recruiting 150 patients completing an 8-month intervention and cohort 2 recruiting 120 patients completing a 6-month intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (18+ years of age)
2. Newly diagnosed patients with lung cancer (non-small cell and small cell lung cancer):

   * Patients with stages I-III lung cancer:

     1) starting multimodality therapy including chemoradiation (either concurrent or sequential), systemic treatment, or radiation alone; and may be followed by surgery; or 2) starting adjuvant therapy after lung resection ((chemotherapy alone, radiation alone, or chemoradiation (either concurrent or sequential))
   * Patients with stage IV lung cancer or recurrent/metastatic:

   Eligible at diagnosis and for up to 3 months after starting treatment

   o Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0-3
3. Vulnerable patients who meet at least one of the following criteria:

   * Economically disadvantaged (household gross monthly income at or below 130% of the Federal Poverty Level)
   * Racial and ethnic minorities (African Americans, American Indians and Alaska Natives, Asians and Pacific Islanders, and Hispanics)
   * No health insurance
   * Elderly patients (ages 65 years or older)
   * Reside in rural areas (non-metropolitan counties with less than 50,000 people)
4. Voluntarily provide consent, HIPPA authorization form, and consent from treating oncologist.
5. Able to speak and read English themselves or with minimal help.
6. Able to receive medically-tailored meals for the course of the study if being assigned to the intervention arm, and willing to sign the MTM agreement.

Exclusion Criteria:

1. Cognitively unable to consent or have physical or mental limitations that would prevent full participation in the program.
2. Have medical conditions that significantly impact digestion, metabolism, or food intake (e.g., surgical loss of esophagus, stomach, or colon; pancreas dysfunction; brain surgery that alters cognition; severe food allergies; etc.) or have active metabolic or digestive illnesses (i.e., Celiac disease, IBS, renal insufficiency, hepatic insufficiency).
3. Pregnant or planning to become pregnant during the study.
4. Unable to receive medically-tailored meals for the course of the study if being assigned to the intervention arm, including lack of a permanent address to which meals can be delivered (a friend or home address is acceptable given it is used on a consistent basis), not having a fully functioning kitchen with a microwave or oven for cooking, not having a standard-sized refrigerator with a freezer with storage capacity to hold one week's worth of meals; or unwilling to sign the MTM agreement.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 299 (Actual)
Dates: Start 2020-11-24 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Nutritional Intake | Baseline, 3-month, and 6 months [for cohort 2] or 8 months [for cohort 1]
  Change in diet quality and intake of key food groups and nutrients as assessed by the National Cancer Institute Diet History Questionnaire (DHQ III)
Weight | Recorded at each clinical visit. From date of beginning baseline until the date of completing the final (6 or 8 month) study visit, an average of 3-4 clinic visits dependent on course of treatment.
  Change in weight measured in the clinic

SECONDARY OUTCOMES:
Food Insecurity | Baseline, 3-month, and 6 months [for cohort 2] or 8 months [for cohort 1]
  Change in food insecurity measured by the U.S. Department of Agriculture (USDA) Household Food Security Survey
Patient-reported Symptoms | Baseline, 3-month, and 6 months [for cohort 2] or 8 months [for cohort 1]
  Change in patient-reported symptoms (fatigue, pain, nausea, vomiting, appetite loss, and sleep disturbance) as assessed by a Patient-Reported Outcomes version of the CTCAE (PRO-CTCAE)
Patient-reported Functional Outcomes - Anxiety | Baseline, 3-month, and 6 months [for cohort 2] or 8 months [for cohort 1]
  Change in patient-reported functional outcomes (physical, social, and cognitive functioning) assessed by General Anxiety Disorder-7 (GAD-7). The total score for the seven items ranges from 0 to 21 (0-4: minimal anxiety. 5-9: mild anxiety. 10-14: moderate anxiety. 15-21: severe anxiety).
Patient-reported Functional Outcomes - Depression | Baseline, 3-month, and 6 months [for cohort 2] or 8 months [for cohort 1]
  Change in patient-reported functional outcomes (physical, social, and cognitive functioning) assessed by Patient Health Questionnaire-9 (PHQ-9). The total score for the nine items ranges from 0 to 27 (0-4: no depression, 5-9: mild depression, 10-14: moderate depression, 15-19: moderately severe depression, 20-27: severe depression).
Health-Related Quality of Life in Cancer Patients | Baseline, 3-month, and 6 months [for cohort 2] or 8 months [for cohort 1]
  Change in quality of life as assessed by the European Organisation for Research and Treatment of Cancer (EORTC) quality of life questionnaire (EORTC-QLQ-30). All of the scales and single-item measures range in score from 0 to100. A high scale score represents a higher response level. Thus a high score for a functional scale represents a high/healthy level of functioning, a high score for the global health status/QoL represents a high QoL, but a high score for a symptom scale/item represents a high level of symptomatology/problems.
Quality of Life in Lung Cancer Patients | Baseline, 3-month, and 6 months [for cohort 2] or 8 months [for cohort 1]
  Change in quality of life as assessed by the European Organisation for Research and Treatment of Cancer (EORTC) quality of life questionnaire lung cancer module (EORTC-QLQ-LC13). All of the scales and single-item measures range in score from 0 to 100. A high score for the scales and single items represents a high level of symptomatology or problems.
Hospitalizations | From baseline until the date of completing the 6 months [for cohort 2] or 8 months [for cohort 1] study visit.
  Rate of hospitalizations will assessed by medical record review and linkage with discharge data
ED visits | From baseline until the date of completing the 6 months [for cohort 2] or 8 months [for cohort 1] study visit.
  Rate of ED visits assessed by medical record review and linkage with discharge data
Treatment-related Toxicities | From baseline until the date of completing the 6 months [for cohort 2] or 8 months [for cohort 1] study visit.
  Rate of treatment-related toxicities assessed by the treating medical oncologist using the National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events (CTCAE)
Treatment Compliance | Recorded at each clinical visit. From date of beginning baseline until the date of completing the final (6 or 8 month) study visit, an average of 3-4 clinic visits dependent on course of treatment.
  Treatment completion (dose reductions and treatment delays) assessed by the treating medical oncologist
Gut Microbial Composition | Baseline, 3-month, and 6 months [for cohort 2] or 8 months [for cohort 1]
  Change in gut microbiome via metagenomic whole shotgun sequencing (mWGS)
Cancer Mortality | 5-8 Years
  National Death Index search performed approximately 5 years after the final patient is enrolled.

OTHER OUTCOMES:
MTM Program Implementation | From consent through study completion, 6 months [for cohort 2] or 8 months [for cohort 1]
  Nutrition counseling adherence (rate of attendance)

CONTACTS AND LOCATIONS:
Overall Officials: FangFang Zhang, MD, PhD, Principal Investigator — Tufts University; Colleen Spees, PhD, MEd, RD, LD, FAND, Principal Investigator — Ohio State University
Locations (4):
- United States (4):
  - Tufts Medical Center, Boston, Massachusetts
  - The James Cancer Hospital, Columbus, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NutriCare Study Website — https://tuftsfoodismedicine.org/project/nutricare/

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-05): https://cdn.clinicaltrials.gov/large-docs/70/NCT04986670/Prot_SAP_001.pdf